CLINICAL TRIAL: NCT04915612
Title: A Phase I Study of Liposomal Cytarabine and Daunorubicin (CPX-351) in Combination With Gemtuzumab Ozogamicin (GO) in Relapsed Refractory Pediatric Patients With Acute Myeloid Leukemia (AML)
Brief Title: Liposomal Cytarabine, Daunorubicin, and Gemtuzumab Ozogamicin for the Treatment of Relapsed Refractory Pediatric Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0484; NCI-2020-13915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0484 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-25; First posted 2021-06-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab; CPX-351; Injections; Daunorubicin; Cytarabine; Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPX-351, GO) (Experimental): INDUCTION 1 (28 days): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.
  INDUCTION 2: Patients who do not attain a defined clinical response after cycle Induction 1 receive CPX-351 IV on days 1 and 3 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Beginning 4 weeks after last induction, patients receive CPX-351 IV over 90 minutes on days 1 and 3 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase I trial studies the best dose and side effects of liposomal cytarabine, daunorubicin, and gemtuzumab ozogamicin in treating pediatric patients with acute myeloid leukemia that has returned after treatment (relapsed) or does not respond to treatment (refractory). Chemotherapy drugs, such as liposomal cytarabine and daunorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to a toxic agent called ozogamicin. Gemtuzumab attaches to CD33 positive cancer cells in a targeted way and delivers ozogamicin to kill them. Giving liposomal cytarabine and daunorubicin and gemtuzumab ozogamicin may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and safety of liposomal cytarabine and daunorubicin (CPX-351) in combination with gemtuzumab ozogamicin (GO) in relapsed refractory pediatric patients with acute myeloid leukemia (AML).

SECONDARY OBJECTIVE:

I. To determine the preliminary assessment of efficacy by overall response (OR), including complete remission (CR), CR with incomplete blood count recovery and partial remission), overall survival (OS), event-free survival (EFS) and duration of response (DOR) of pediatric patients treated with this combination.

EXPLORATORY OBJECTIVES:

I. To determine the minimal residual disease (MRD) after treatment with this combination and its impact in long-term outcome (OS and EFS).

II. To determine the effect of the level of pre-treatment expression of CD33 with response to this combination.

III. To determine the effect of this treatment combination on responding pediatric patients transitioning to hematopoietic stem cell transplant (HSCT) i.e., number and percentage of patients that are able to transition to HSCT.

OUTLINE:

INDUCTION 1 (28 days): Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.

INDUCTION 2: Patients who do not attain a defined clinical response after cycle Induction 1 receive CPX-351 IV on days 1 and 3 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Beginning 4 weeks after last induction, patients receive CPX-351 IV over 90 minutes on days 1 and 3 and GO IV over 2 hours on day 1 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with diagnosis of CD33 positive (> 3%),

  * Newly diagnosed secondary AML
  * Relapsed refractory acute myeloid leukemia by World Health Organization (WHO) criteria Patients must have >= 5% blasts in the bone marrow as assessed by morphology or flow cytometry. However, if an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia with >= 5% blasts in the peripheral blood
* Pediatric Patients with myelodysplastic syndrome (MDS) who progress to AML are eligible at the time of diagnosis of AML regardless of any prior therapy for MDS
* Performance status: Lansky >= 50 for patients who are =< 16 years old and Karnofsky >= 50% for patients who are > 16 years old
* Age =< 21 years of age
* Total serum bilirubin =< 2 x upper limit of normal (ULN). Patients with known Gilbert's syndrome may have a total bilirubin up to =< 3 x ULN
* Serum creatinine =< 2.0 mg/dl
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 3 x ULN; =< 5 x ULN in case of suspected leukemic liver involvement
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug. Effective methods of birth control include:

  * Birth control pills, skin patches, shots, implants (placed under the skin by a health care provider)
  * Intrauterine devices (IUDs)
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with Spermicide
  * Abstinence
* Males, need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 30 days after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 30 days after the last treatment

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated and in remission. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses)
* Presence of clinically significant uncontrolled central nervous system (CNS) pathology such as epilepsy, childhood seizure, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis
* Evidence of active cerebral/meningeal disease. Patients may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of consent with at least 2 consecutive spinal fluid negative assessments for residual leukemia and negative imaging (imaging required only if previously showing evidence of CNS leukemia not otherwise documented by spinal fluid assessment)
* Patients with a cardiac ejection fraction (as measured by either multigated acquisition scan [MUGA] or echocardiogram) < 50% are excluded
* Patients with total cumulative doses of non-liposomal daunorubicin, or other anthracycline equivalent, greater than 450 mg/m^2
* Patients with uncontrolled, active infections (viral, bacterial, or fungal). Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable
* Known active hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Liver cirrhosis or other serious active liver disease or with suspected active alcohol abuse
* Active acute/chronic graft-versus-host disease (GvHD) requiring systemic treatment; or receiving immunosuppression for GvHD prophylaxis within 2 weeks from the start of study therapy
* Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exception:

  * To reduce the circulating blast count or palliation: Single dose intravenous cytarabine or hydroxyurea. No washout necessary for these agents
* Females who are pregnant or lactating
* Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards
* Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, or bone marrow failure syndromes are not eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days
  Will employ the Bayesian optimal interval (BOIN) design.
Incidence of adverse events | Up to 28 days
  The overall incidence and severity of all adverse events using Common Toxicity Criteria version 4.0.

SECONDARY OUTCOMES:
Objective response | Up to 28 days
  Will be summarized using descriptive statistics overall and per dose levels.
Duration of response | Number of days from the date of initial response (partial response or better) to the date of first documented disease progression/relapse or death, whichever occurs first, assessed p to 28 days
  Will be summarized using descriptive statistics overall and per dose levels.
Overall survival | Number of days from study enrollment to death due to any cause, assessed up to 28 days
  Will be estimated using Kaplan-Meier method.
Event free survival | Number of days from the date of treatment initiation to the date of documented treatment failure, relapses from complete response, or death from any cause, whichever occurs first, assessed up to 28 days
  Will be estimated using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Branko Cuglievan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04915612/ICF_000.pdf